CLINICAL TRIAL: NCT00936559
Title: Randomized, Single-Blind, Standard Of Care Control, Dose-Escalating, Multicenter, Safety Study Of BMP-655/ACS As An Adjuvant Therapy For Treatment Of Full Thickness Rotator Cuff Tears Treated By Means Of An Open Surgical Procedure
Brief Title: Study Evaluating Safety Of BMP-655/ACS As An Adjuvant Therapy For Rotator Cuff Repair
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 3202V1-1001
Record Dates: First submitted 2009-07-02; First posted 2009-07-10 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Rotator Cuff Tear
Keywords: rotator cuff tear repair; open surgical technique; safety
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Arm A
  Interventions: Biological: BMP-655/ACS or Standard of Care
- 2 (Experimental): Arm B
  Interventions: Biological: BMP-655/ACS or Standard of Care
- 3 (Experimental): Arm C
  Interventions: Biological: BMP-655/ACS or Standard of Care

INTERVENTIONS:
Biological: BMP-655/ACS or Standard of Care — Decision was made by Legal to withhold this information
  Arms: 1
Biological: BMP-655/ACS or Standard of Care — Decision was made by Legal to withhold this information.
  Arms: 2
Biological: BMP-655/ACS or Standard of Care — Decision was made by Legal to withhold this information,
  Arms: 3

SUMMARY:
Study to assess the safety of 3 differing concentrations of BMP-655/ACS in subjects with full thickness Rotator Cuff Tears (RCTs).

DETAILED DESCRIPTION:
This decision to terminate enrollment in this study is based on the company's change in prioritization for the portfolio and was not due to any safety concerns, or regulatory interactions.

Patients already enrolled in the study, should continue to complete assessments as described in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects and surgically sterile or postmenopausal female subjects between the ages of 25 and 75 years old with specific full-thickness RCTs identified on closed MRI within 3 months before surgery.

Exclusion Criteria:

* Subjects who have had previous surgical intervention to the shoulder joint under study or additional injury requiring surgical repair or a history of shoulder dislocation in the affected shoulder or physical examination findings of instability in either shoulder
* Subjects who are unable to complete functional evaluations because of any other concurrent injuries or impairment in either the arm
* Subjects identified with specific fatty infiltration of their RC muscles on MRI taken within 3 months prior to surgical repair
* Subjects with moderate or severe degenerative arthritis of the shoulder under study or any bone abnormalities as confirmed on a radiograph
* Subjects with rheumatologic conditions affecting the shoulder joints or autoimmune disorders, treated with more than 3 corticosteroid injections in the shoulder under study within 1 year of planned surgery, any recent corticosteroid injection in the shoulder or currently receiving oral corticosteroids
* Subjects who are either unwilling or unable to undergo examination with closed MRI.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Abnormal X-rays, MRIs, CT scans, physical examination of limb, functional evaluations, AE/SAE, vital signs, subject assessment of pain, lab tests | 1 year

SECONDARY OUTCOMES:
Investigator Questionnaire | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Germany (2):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Hamburg
- Netherlands (2):
  - Pfizer Investigational Site, Amsterdam
  - Pfizer Investigational Site, Hoofddorp

REFERENCES:
- [Derived] Ide J, Mochizuki Y, van Noort A, Ochi H, Sridharan S, Itoi E, Greiner S. Local rhBMP-12 on an Absorbable Collagen Sponge as an Adjuvant Therapy for Rotator Cuff Repair-A Phase 1, Randomized, Standard of Care Control, Multicenter Study: Part 2-A Pilot Study of Functional Recovery and Structural Outcomes. Orthop J Sports Med. 2017 Sep 12;5(9):2325967117726740. doi: 10.1177/2325967117726740. eCollection 2017 Sep. PMID 28932752
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3202V1-1001&StudyName=Study%20Evaluating%20Safety%20Of%20BMP-655/ACS%20As%20An%20Adjuvant%20Therapy%20For%20Rotator%20Cuff%20Repair